CLINICAL TRIAL: NCT05544500
Title: Immediate and Residual Effects of Functional Chewing Gum on Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Perfetti van Melle SPA (Unknown)
Responsible Party: Principal Investigator, Crystal Haskell-Ramsay, Professor, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 63O2
Record Dates: First submitted 2022-09-08; First posted 2022-09-16 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, counterbalanced crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Sugar-free tablet
  Interventions: Dietary Supplement: Placebo
- Basic sugar-free gum (Active Comparator): Sugar-free chewing gum
  Interventions: Dietary Supplement: Basic Chewing Gum
- Functional gum (Experimental): Sugar-free chewing gum with functional ingredients
  Interventions: Dietary Supplement: Functional Gum

INTERVENTIONS:
Dietary Supplement: Functional Gum — Functional gum containing a proprietary composition of a herbal extract and vitamins
  Arms: Functional gum
Dietary Supplement: Basic Chewing Gum — Sugar-free chewing gum
  Arms: Basic sugar-free gum
Dietary Supplement: Placebo — Sugar-free tablet
  Arms: Placebo

SUMMARY:
Previous research suggests that chewing gum may influence several functions including attention and alertness. Gum can also be used as a vehicle for delivering ingredients that have the ability to modulate attention and mood. This study will explore the effects of a functional gum containing a proprietary composition of a herbal extract and vitamins. These effects will be compared to the effects of a basic sugar-free gum and to a tablet which will include the same ingredients as the basic sugar-free gum. Effects will be explored on computerised measures of attention/concentration and via ratings of current mood. The study will assess the immediate effects of chewing gum as well as the effects 1 hour later.

There will be an initial remote screening session followed by visits to the laboratory on 4 separate occasions: an introductory/training visit and three active study days.

DETAILED DESCRIPTION:
This randomised, double-blind, placebo-controlled, counterbalanced crossover study will assess the acute effects of chewing functional gum on measures of concentration and mental acuity in healthy participants in comparison to basic sugar free gum and placebo.

The trial will utilise the COMPASS cognitive assessment system and a series of subjective mood measures. The core cognitive assessment of study will employ a selection of tasks assessing performance within the 'Psychomotor Speed', 'Sustained Attention', and 'Decision Making' cognitive domains. Subjective changes in mood ('alertness', 'stress', 'tranquillity', concentration', 'focus' and 'mental tiredness') will also be assessed.

Assessments will take place at baseline, during treatment consumption and 1 hour post-dose to assess the residual effects following chewing.

Participants will have an initial remote screening session followed by visits to the laboratory on 4 separate occasions: an introductory/training visit (Day 0) and three active study days (Day 1, Day 2, and Day 3) spaced 2 days apart (+5 days).

The remote screening session will be completed via telephone call and will comprise: briefing on requirements of the study, obtaining of informed consent via completion of an online consent form, health screening, collection of demographic data, and completion of the Caffeine Consumption Questionnaire (CCQ).

The introductory/training visit to the laboratory will begin with physiological eligibility measures that cannot be completed remotely (e.g. height and weight, waist-to-hip ratio) followed by training on the cognitive and mood measures.

Following the introductory visit participants will attend the laboratory at either 10 am or 2 pm on three separate occasions (Day 1, Day 2, and Day 3) with testing time consistent within participants and counterbalanced across treatment orders. All testing days (will be identical, with the exception that the participants will consume a different treatment at each visit.

On each testing visit participants will be required to eat a standard meal at least 1 hour before testing and to abstain from alcohol and over the counter medications (including hay fever medications) for 24 hours and caffeinated products for 5 hours before testing (meal items should be kept consistent across visits). Participants will arrive to the laboratory at their allotted time and, following completion of the Case Report Form (to confirm continued compliance with inclusion/exclusion criteria), complete a baseline assessment for that day (10 mins). They will then be randomised to treatment order (Day 1 only). Participants will have a 10-minute rest before completing the tasks again whilst 'chewing' their allotted treatment for that day (10 mins). Following this they will dispose of their treatment and then complete a final assessment 1 hour later to assess the residual effects following chewing.

Testing will take place in a suite of testing facilities with participants visually isolated from each other.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health
* Aged 18 to 35 years at the time of giving consent
* Report good oral health and chewing ability
* Proficient in English

Exclusion Criteria:

* Have any pre-existing medical condition/illness which will impact taking part in the study NOTE: There may be unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance.
* Are currently taking prescription medications NOTE: the explicit exception to this are contraceptive treatments for female participants, topical skin treatments e.g. for eczema, acne, and those taken 'as needed' in the treatment of hay fever. As above, there may be other instances of medication use which, where no interaction with the active treatments is likely, and which would not be expected to have any impact on brain function, participants may be able to progress to screening. Use of any medications which impact mood or cognitive function e.g. anti depressants, anti anxiety medications etc. are not permitted.
* Have undergone dental treatment 1 week before the test, or needs or is planning dental treatments during the study (excluding routine dental check-up)
* Have a Body Mass Index (BMI) outside of the range 18.5-30 kg/m2
* Are pregnant, seeking to become pregnant or lactating.
* Have a visual impairment that cannot be corrected with glasses or contact lenses (excluding colour-blindness)
* Smoke tobacco or vape nicotine or use nicotine replacement products (occasional social smoking is permitted)
* Have relevant food intolerances/ sensitivities/ allergies
* Have taken dietary supplements e.g. Vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement washout prior to participating and for the duration of the study on the proviso that the supplements are taken are out of choice and are not medically prescribed or advised). Existing and consistent use of vitamin D supplements and protein shakes are permitted
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Simple Reaction Time | During treatment consumption, adjusted for baseline
  Cognitive Function - attention
Choice Reaction Time | During treatment consumption, adjusted for baseline
  Cognitive Function - attention
Digit Vigilance | During treatment consumption, adjusted for baseline
  Cognitive Function - attention
Simple Reaction Time | 1-hour post-consumption, adjusted for baseline
  Cognitive Function - attention
Choice Reaction Time | 1-hour post-consumption, adjusted for baseline
  Cognitive Function - attention
Digit Vigilance | 1-hour post-consumption, adjusted for baseline
  Cognitive Function - attention

SECONDARY OUTCOMES:
COMPASS VAMS (Visual Analogue Mood Scales) | During treatment consumption, adjusted for baseline
  Mood
Concentration VAS (Visual Analogue Scale) | During treatment consumption, adjusted for baseline
  Mood
Focused VAS (Visual Analogue Scale) | During treatment consumption, adjusted for baseline
  Mood
Mentally tired VAS (Visual Analogue Scale) | During treatment consumption, adjusted for baseline
  Mood
COMPASS VAMS (Visual Analogue Mood Scales) | 1-hour post-consumption, adjusted for baseline
  Mood
Concentration VAS (Visual Analogue Scale) | 1-hour post-consumption, adjusted for baseline
  Mood
Focused VAS (Visual Analogue Scale) | 1-hour post-consumption, adjusted for baseline
  Mood
Mentally tired VAS (Visual Analogue Scale) | 1-hour post-consumption, adjusted for baseline
  Mood

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell-Ramsay, Principal Investigator — Northumbria University
Locations (1):
- Department of Psychology, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haworth E, Haskell-Ramsay CF. Immediate and residual effects of functional chewing gum on sustained attention and mood. Nutr Neurosci. 2025 Apr;28(4):439-447. doi: 10.1080/1028415X.2024.2379698. Epub 2024 Jul 23. PMID 39039933